CLINICAL TRIAL: NCT03067103
Title: Comparison of Effect of Peritonsillar Infiltration of Ketamine and Tramadol on Pediatric Posttonsillectomy Pain: A Double-blinded Randomized Placebo-controlled Clinical Trial
Brief Title: Comparison of Peritonsillar Infiltration of Tramadol Ketamine and Placebo on Pediatric Posttonsillectomy Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, juliana alves de sousa caixeta, Medical assistant, Universidade Federal de Goias
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: JASC1; 48547215.0.0000.5076 (Other: intitution's Ehtical approval)
Record Dates: First submitted 2017-02-12; First posted 2017-03-01 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Sleep Disorder; Breathing-Related; Pain, Postoperative; Child, Only
Keywords: Adenotonsillectomy; pain; topic analgesia; child
MeSH Terms: conditions — Sleep Wake Disorders; Pain, Postoperative; Pain | interventions — Tramadol; Ketamine

STUDY DESIGN:
Intervention Model Description: Patientes will be seleted to receive peritonsillar injection of Tramadol, Ketamine or Placebo before tonsillectomy prospective, double-blind, placebo controlles
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients admitted for tonsillectomy were randomized into 3 groups by means of sealed envelopes. The envelope selected by the caregiver will be open by the registered nurse, who will prepare the infiltration. Neither the surgeon, anesthesiologist the caregiver nor the patient will see what is inside the envelope. The register of the envelope number and patient data will be done by the statistical group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tramadol (Active Comparator): Tramadol group will receive 2 mg/kg (2 ml) through the peritonsillar fossa. For each tonsil 1 ml will be applied to upper pole, lower pole and between the upper and lower pole with 25-G needle. The depth of the infiltration will be as superficial as 3 mm of needle injected and ballooned out the submucosal tissues of the tonsillar pillar, intratonsillar injection as avoided.
  Interventions: Drug: Tramadol
- ketamine (Active Comparator): Ketamine group will receive 0.5 mg/kg (2cc) through the peritonsillar fossa. For each tonsil 1 ml will be applied to upper pole, lower pole and between the upper and lower pole with 25-G needle. The depth of the infiltration will be as superficial as 3 mm of needle injected and ballooned out the submucosal tissues of the tonsillar pillar, intratonsillar injection as avoided.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Placebo group will receive 2mL of saline solution through the peritonsillar fossa. For each tonsil 1 ml will be applied to upper pole, lower pole and between the upper and lower pole with 25-G needle. The depth of the infiltration will be as superficial as 3 mm of needle injected and ballooned out the submucosal tissues of the tonsillar pillar, intratonsillar injection as avoided.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Tramadol — Patients will receive injections in peritonsillar fossa of tramadol (2 mg/kg-2 ml)
  Other Names: group 1
  Arms: tramadol
Drug: Ketamine — Patients will receive injections in peritonsillar fossa of ketamine prior to surgery
  Other Names: Group 2
  Arms: ketamine
Drug: Placebos — Patients will receive 2mL of saline solution in peritonsillar fossa prior to surgery
  Other Names: Group 3
  Arms: Placebo

SUMMARY:
Adenotonsillectomy is one of the most common ambulatory surgical procedures performed to children. Tonsillectomy or adenotonsillectomy have a high incidence of postoperative pain. There is still debate about the optimal analgesia for this common surgical procedure. Different methods have been described and used to reduce pain including; improved intraoperative anesthetic pain regimens, use of corticosteroids, adjustment of surgical technique, and intraoperative local anesthetic injection. Intraoperative local anesthetic is a preventive or preemptive analgesia which is the analgesia given before painful stimuli to prevent the subsequent pain. The main goal of the preventive analgesia is the pain relief with minimum side effects. The role of local anesthetic infiltration in the reduction of postadenotonsillectomy pain is still controversial. The objective of this study is to investigate and compare the effectiveness of preincisional peritonsillar infiltration of ketamine and tramadol for post-operative pain on children following adenotonsillectomy. This is prospective, double-blinded randomized study.

DETAILED DESCRIPTION:
Adenotonsillectomy is one of the most common ambulatory surgical procedures performed to children. Tonsillectomy or adenotonsillectomy have a high incidence of postoperative pain. There is still debate about the optimal analgesia for this common surgical procedure. Different methods have been described and used to reduce pain including. The main goal of the preventive analgesia is the pain relief with minimum side effects. The role of local anesthetic infiltration in the reduction of postadenotonsillectomy pain is still controversial. Blockage of N-methyl-D-aspartate (NMDA) activation and interception of nociceptive in put are important factors to achieve the reduction in subsequent pain. Ketamine hydrochloride is an NMDA receptor antagonist. The blockage of the NMDA channel and analgesic properties are both at subanesthetic doses for the ketamine. Ketamine also prevents central sensitization of nociceptors. Previous studies described the analgesic effect of intravenous application or peritonsillar infiltration of ketamine intraoperatively in children after tonsillectomy. Tramadol is another analgesic and a synthetic opioid of the aminocyclohexanol group which is a central opioid agonist with less respiratory depression compared to morphine. We knew that tramadol has both systemic and local anesthetic effect on peripheral nerves from human and animal studies.

The study was approved by the Ethics Committee of the University. The consents will be taken from all parents. Patients will be randomized from seald envelope into tramadol, ketamine or control (serum physiologic) to receive the preincisional peritonsillar infiltration before the surgery. There will de 36 patients in each group. The study drug is supplied of a liquid identical in color and volume. All surgeons, anesthesiologists, nurses, patients and parents will be blinded to study group until the end of the study All children will receive a premedication including midazolam hydrochloride (0.5 mg/kg; maximum dose, 20 mg) followed by a standard general inhalational anesthetic (50% O2-N2O and 8% sevoflurane). Children also received 0.1 mg/kg of fentanyl citrate and 0.2 mg/kg mivacurium intravenously. After the intubation maintenance anesthesia will be keep with nitrous oxide (50%) in oxygen and sevoflurane. All patients will receive the peritonsillar injection of the study drug before the excision of the anesthesia. Tramadol group will receive 2 mg/kg (2 ml), ketamine group 0.5 mg/kg (2cc), control group 2 ml of serum physiologic. All infiltrations will be through the peritonsillar fossa. For each tonsil 1 ml will be applied to upper pole, lower pole and between the upper and lower pole with 25-G needle. After the infiltration surgeons will wait 3 min for tonsillectomy. The same standard blunt dissection will be performed to all children by the same surgeon. During the operation heart rate oxygen saturation, average blood pressure, respiration rates will be recorded in every 5 min. Operation, anesthesia times will also be recorded. Postoperatively pain, nausea, vomiting, sedation scores, the existence of dysphagia, bleeding were recorded at 2, 6, 12, 24 h postoperatively. Children's pain scores will be measured by using Visual Analogue Scale (VAS).If the pain score is greater than 5, Ibuprofen will be given to children. Pains with the request for analgesic requirements, the time of analgesia requirement, patient satisfaction will be also recorded.

Data analysis will be performed by using SPSS for Windows. The relationship between categorical variables will be test by Chi-square test and Anova test will be performed to compare groups according to continuous variables. Also LSD test will be used to detect subgroup differences. p Values higher than 0.05 will be considered as significant. Mean and standard deviations and percentages will be given as descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Sleep disordered breathing
* ASA I-II

Exclusion Criteria:

* ASA III-IV physical status
* Coagulation disturbances
* Presence of relevant drug allergies
* pulmonary and cardiac diseases
* Craniofacial anomalies
* Mental diseases
* Genetic disorders
* Peritonsillar abscess formation
* Regular use of analgesics 24 h prior to surgery

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2017-07-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Peritonsillar infiltration of ketamine reduces postoperative pain in children undergone adenotonsillectomy | 24h
  Children will be evaluated by the Visual Analog Scale of pain and children who had received ketamine should be lower scores when compared to children who had received placebo. These children are expected to ask less times for analgesic medication;

SECONDARY OUTCOMES:
Peritonsillar infiltration of tramadol reduces postoperative pain in children undergone | 24h
  Children will be evaluated by the Visual Analog Scale of pain and children who had received tramadol should be lower scores when compared to children who had received placebo. These children are expected to ask less times for analgesic medication;

CONTACTS AND LOCATIONS:
Overall Officials: juliana a caixeta, MD, Principal Investigator — Assistant Doctor
Locations (1):
- Juliana Alves de Sousa Caixeta, Anápolis, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ugur KS, Karabayirli S, Demircioglu RI, Ark N, Kurtaran H, Muslu B, Sert H. The comparison of preincisional peritonsillar infiltration of ketamine and tramadol for postoperative pain relief on children following adenotonsillectomy. Int J Pediatr Otorhinolaryngol. 2013 Nov;77(11):1825-9. doi: 10.1016/j.ijporl.2013.08.018. Epub 2013 Aug 27. PMID 24041860
- [Background] Yenigun A, Et T, Aytac S, Olcay B. Comparison of different administration of ketamine and intravenous tramadol hydrochloride for postoperative pain relief and sedation after pediatric tonsillectomy. J Craniofac Surg. 2015 Jan;26(1):e21-4. doi: 10.1097/SCS.0000000000001250. PMID 25569408
- [Background] Ayatollahi V, Behdad S, Hatami M, Moshtaghiun H, Baghianimoghadam B. Comparison of peritonsillar infiltration effects of ketamine and tramadol on post tonsillectomy pain: a double-blinded randomized placebo-controlled clinical trial. Croat Med J. 2012 Apr;53(2):155-61. doi: 10.3325/cmj.2012.53.155. PMID 22522994
- [Background] Heiba MH, Atef A, Mosleh M, Mohamed R, El-Hamamsy M. Comparison of peritonsillar infiltration of tramadol and lidocaine for the relief of post-tonsillectomy pain. J Laryngol Otol. 2012 Nov;126(11):1138-41. doi: 10.1017/S0022215112002058. Epub 2012 Sep 19. PMID 22989763
- [Background] Tong Y, Ding XB, Wang X, Ren H, Chen ZX, Li Q. Ketamine peritonsillar infiltration during tonsillectomy in pediatric patients: An updated meta-analysis. Int J Pediatr Otorhinolaryngol. 2014 Oct;78(10):1735-41. doi: 10.1016/j.ijporl.2014.07.036. Epub 2014 Aug 1. PMID 25139134
- [Background] Siddiqui AS, Raees US, Siddiqui SZ, Raza SA. Efficacy of pre-incisional peritonsillar infiltration of ketamine for post-tonsillectomy analgesia in children. J Coll Physicians Surg Pak. 2013 Aug;23(8):533-7. PMID 23930866
- [Background] Beigh Z, Ul Islam M, Ahmad S, Ahmad Pampori R. Effects of Peritonsillar Injection of Tramadol and Adrenaline before Tonsillectomy. Iran J Otorhinolaryngol. 2013 Jun;25(72):135-40. PMID 24303433